CLINICAL TRIAL: NCT02025400
Title: Phase I Study Comparing Internet Delivered Home Exercise Programs to Standard Orthopedic Care and Outpatient Physical Therapy.
Brief Title: Internet Enhanced, Patient-Centered Orthopedic Care: A Prospective, Randomized, Controlled Pilot Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charlotte Sports Medicine Institute, PA (Other)
Collaborators: Advanced Orthopedic Specialists (Unknown); The Orthopaedic Center (Unknown)
Responsible Party: Principal Investigator, Jonathan Paul, MD, Director, Charlotte Sports Medicine Institute, PA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eRehab101
Record Dates: First submitted 2013-12-26; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Knee Injuries; Shoulder Injuries; Rotator Cuff Disease; Meniscus Tear; Patellofemoral Pain
Keywords: Rehabilitation; eRehab; Physical Therapy; e-Health; Telemedicine; Telerehabilitation; Patient-Centered
MeSH Terms: conditions — Knee Injuries; Shoulder Injuries; Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Therapy (Active Comparator): This arm will receive the standard of care for orthopedic patients receiving a diagnosis and then a recommendation for outpatient physical therapy referral. They will follow through on the referral and attend physical therapy.
  Interventions: Other: Formal Physical Therapy
- eRehab (Experimental): This group will not go to formal therapy but receive Internet delivered patient education and exercise instruction. This group will then perform those exercises at home.
  Interventions: Other: eRehab

INTERVENTIONS:
Other: eRehab — Growth in e-Health applications, defined as any computer or Internet application integrated into health services, has resulted in the development of treatment strategies to improve healthcare while reducing costs. The utilization of e-Health to provide a rehabilitative intervention has recently been identified in the cardiac literature as "e-rehabilitation" or "eRehab." This study specifically compares an orthopedic eRehab Internet application to standard outpatient physical therapy as an adjunct in the treatment of non-complicated knee and shoulder disorders.
  Arms: eRehab
Other: Formal Physical Therapy — This intervention involves referral to a licensed physical therapist or supervised ATC-L.
  Arms: Physical Therapy

SUMMARY:
The investigators have previously reported on patient utilization of an eRehab patient education web portal that utilizes streaming, clinician prescribed video instruction to motivate and inform patients in self-care of their orthopedic condition, focusing on the importance of a home exercise program. The greatest barrier to patient use of this web-based home exercise treatment plan was the initial access to the program. The purpose of this study is to compare an Internet-based patient education rehab portal (eRehab) to formal physical therapy (PT) in terms of patient costs and outcomes.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled pilot study. Twenty-four patients who were candidates for a knee or shoulder orthopedic outpatient physical therapy referral were randomized to a 6-week treatment course of either PT or eRehab. Patients were evaluated for outcome scores (KOOS or DASH), pain NRS-11 scores, patient subjective outcomes and cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed by board certified orthopedic surgeon to be in need of formal physical therapy referral
* had the ability to access and use the Internet and email
* English-speaking
* non-pregnant adults
* had not received formal physical therapy for their current diagnosis

Exclusion Criteria:

* work-related injuries
* pain NRS-11 score greater than or equal to 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Outcome scores for knee (KOOS) and shoulder (DASH) | six weeks

SECONDARY OUTCOMES:
NRS-11 pain scores | 6 weeks

OTHER OUTCOMES:
Patient utilization of an eRehab portal measured by number of logons and performance of a home exercise program as documented with an exercise log. | 6 weeks
Patient cost of care per episode | 6 months
  A patient's insurance explanation of benefits will be reviewed for 6 months from completion of the current episode of care to determine patient out of pocket expenses
Total cost of care per episode | 6 months
  Each patient's EOB will be reviewed to determine total cost of care for each episode of care

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Orthopaedic Specialists, Prince Frederick, Maryland
  - Charlotte Sports Medicine Institute, Charlotte, North Carolina

REFERENCES:
- [Background] Burden of Musculoskeletal Diseases in the United States: Prevalence, Societal and Economic Cost. Rosemont, IL, American Academy of Orthopaedic Surgeons. February 2008.
- [Background] Eng TR. The eHealth Landscape: A Terrain Map of Emerging Information and Communication Technologies in Health and Health Care. Princeton, NJ: The Robert Wood Johnson Foundation, 2001.
- [Result] Antypas K, Wangberg SC. E-Rehabilitation - an Internet and mobile phone based tailored intervention to enhance self-management of cardiovascular disease: study protocol for a randomized controlled trial. BMC Cardiovasc Disord. 2012 Jul 9;12:50. doi: 10.1186/1471-2261-12-50. PMID 22776554
- [Result] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269
- [Result] APTA Presentation to House Ways and Means Committee, 2011
- [Result] Farley FA, Weinstein SL. The case for patient-centered care in orthopaedics. J Am Acad Orthop Surg. 2006 Aug;14(8):447-51. doi: 10.5435/00124635-200608000-00001. PMID 16885475
- [Result] Fatehi F, Wootton R. Telemedicine, telehealth or e-health? A bibliometric analysis of the trends in the use of these terms. J Telemed Telecare. 2012 Dec;18(8):460-4. doi: 10.1258/jtt.2012.gth108. Epub 2012 Dec 3. PMID 23209265
- [Result] Galea MP, Levinger P, Lythgo N, Cimoli C, Weller R, Tully E, McMeeken J, Westh R. A targeted home- and center-based exercise program for people after total hip replacement: a randomized clinical trial. Arch Phys Med Rehabil. 2008 Aug;89(8):1442-7. doi: 10.1016/j.apmr.2007.11.058. Epub 2008 Jun 30. PMID 18586222
- [Result] Grant JA, Mohtadi NG, Maitland ME, Zernicke RF. Comparison of home versus physical therapy-supervised rehabilitation programs after anterior cruciate ligament reconstruction: a randomized clinical trial. Am J Sports Med. 2005 Sep;33(9):1288-97. doi: 10.1177/0363546504273051. Epub 2005 Jul 7. PMID 16002493
- [Result] Russell TG, Buttrum P, Wootton R, Jull GA. Internet-based outpatient telerehabilitation for patients following total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2011 Jan 19;93(2):113-20. doi: 10.2106/JBJS.I.01375. PMID 21248209
- [Result] Helwig AL, Lovelle A, Guse CE, Gottlieb MS. An office-based Internet patient education system: a pilot study. J Fam Pract. 1999 Feb;48(2):123-7. PMID 10037543
- [Result] Hill AM, McPhail S, Hoffmann T, Hill K, Oliver D, Beer C, Brauer S, Haines TP. A randomized trial comparing digital video disc with written delivery of falls prevention education for older patients in hospital. J Am Geriatr Soc. 2009 Aug;57(8):1458-63. doi: 10.1111/j.1532-5415.2009.02346.x. Epub 2009 Jun 8. PMID 19515102
- [Result] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Result] Jolly K, Taylor R, Lip GY, Greenfield S, Raftery J, Mant J, Lane D, Jones M, Lee KW, Stevens A. The Birmingham Rehabilitation Uptake Maximisation Study (BRUM). Home-based compared with hospital-based cardiac rehabilitation in a multi-ethnic population: cost-effectiveness and patient adherence. Health Technol Assess. 2007 Sep;11(35):1-118. doi: 10.3310/hta11350. PMID 17767899
- [Result] Ko V, Naylor J, Harris I, Crosbie J, Yeo A, Mittal R. One-to-one therapy is not superior to group or home-based therapy after total knee arthroplasty: a randomized, superiority trial. J Bone Joint Surg Am. 2013 Nov 6;95(21):1942-9. doi: 10.2106/JBJS.L.00964. PMID 24196464
- [Result] Kuhn JE. Exercise in the treatment of rotator cuff impingement: a systematic review and a synthesized evidence-based rehabilitation protocol. J Shoulder Elbow Surg. 2009 Jan-Feb;18(1):138-60. doi: 10.1016/j.jse.2008.06.004. Epub 2008 Oct 2. PMID 18835532
- [Result] Mazzuca SA, Brandt KD, Katz BP, Dittus RS, Freund DA, Lubitz R, Hawker G, Eckert G. Comparison of general internists, family physicians, and rheumatologists managing patients with symptoms of osteoarthritis of the knee. Arthritis Care Res. 1997 Oct;10(5):289-99. doi: 10.1002/art.1790100503. PMID 9362595
- [Result] McCarthy CJ, Mills PM, Pullen R, Richardson G, Hawkins N, Roberts CR, Silman AJ, Oldham JA. Supplementation of a home-based exercise programme with a class-based programme for people with osteoarthritis of the knees: a randomised controlled trial and health economic analysis. Health Technol Assess. 2004 Nov;8(46):iii-iv, 1-61. doi: 10.3310/hta8460. PMID 15527668
- [Result] Paul JJ, Rolfes K, Herron B, Rouse J. Orthopedic eRehab: An Assessment of Patient Utilization of Internet-based Home Exercise Programs. Submitted to Am J Sports Med.
- [Result] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Result] Rozental TD, Bozentka DJ, Beredjiklian PK. Patient education through the Internet: academic and private practice sites. Clin Orthop Relat Res. 2004 Apr;(421):50-3. PMID 15123925
- [Result] Simek EM, McPhate L, Haines TP. Adherence to and efficacy of home exercise programs to prevent falls: a systematic review and meta-analysis of the impact of exercise program characteristics. Prev Med. 2012 Oct;55(4):262-275. doi: 10.1016/j.ypmed.2012.07.007. Epub 2012 Jul 17. PMID 22813920
- [Result] Tunay VB, Baltaci G, Atay AO. Hospital-based versus home-based proprioceptive and strengthening exercise programs in knee osteoarthritis. Acta Orthop Traumatol Turc. 2010;44(4):270-7. doi: 10.3944/AOTT.2010.2306. PMID 21252603
- [Result] Veroff DR, Sullivan LA, Shoptaw EJ, Venator B, Ochoa-Arvelo T, Baxter JR, Manocchia M, Wennberg D. Improving self-care for heart failure for seniors: the impact of video and written education and decision aids. Popul Health Manag. 2012 Feb;15(1):37-45. doi: 10.1089/pop.2011.0019. Epub 2011 Oct 17. PMID 22004181